CLINICAL TRIAL: NCT00918203
Title: A Randomized Phase 2 Study of Human Anti-PDGFRα Monoclonal Antibody (IMC-3G3) With Paclitaxel/Carboplatin or Paclitaxel/Carboplatin Alone in Previously Untreated Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Paclitaxel/Carboplatin With or Without Olaratumab (IMC-3G3) in Previously Untreated Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13900; CP15-0804 (Other: ImClone Systems); I5B-IE-JGDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung neoplasms; IMC-3G3; carboplatin; paclitaxel; PDGFr
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — olaratumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel + Carboplatin (Active Comparator): (Initial 4-6 cycles) Paclitaxel 200 milligram/square meter (mg/m2) over 3 hrs (Day 1) Carboplatin Area Under Concentration (AUC)=6 (Day 1) of each 21-day cycle (Initial 4-6 cycles) Paclitaxel 200 mg/m2 over 3 hrs (Day 1) Carboplatin AUC=6 (Day 1) of each 21-day cycle
  Participants who experience progressive disease may cross over to olaratumab monotherapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Olaratumab + Paclitaxel + Carboplatin (Experimental): (Initial 4-6 cycles)
  Olaratumab 15 milligrams/kilogram (mg/kg) over 30 mins (Days 1 and 8) plus Paclitaxel 200 mg/m2 over 3 hrs (Day 1) Carboplatin AUC=6 (Day 1) of each 21-day cycle
  Participants can remain on study after completing chemotherapy and receive olaratumab monotherapy on Days 1 and 8, provided there is ongoing evidence of clinical benefit.
  Interventions: Biological: Olaratumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Olaratumab — 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, administered intravenously (IV) at 25 milligram/minute (mg/min), with a minimum infusion time of 30 minutes.
  Other Names: LY3012207; IMC-3G3
  Arms: Olaratumab + Paclitaxel + Carboplatin
Drug: Paclitaxel — 200 mg/m2 is then administered IV over 3 hours
Drug: Carboplatin — AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.

SUMMARY:
The purpose of this study is to determine if participants with untreated locally advanced or metastatic non-small cell lung cancer have a better outcome when treated with olaratumab in combination with paclitaxel/carboplatin then when treated with paclitaxel/carboplatin alone.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the progression-free survival (PFS) in previously untreated participants with Stage IIIB/IV non-small cell lung cancer (NSCLC) treated with olaratumab plus paclitaxel and carboplatin versus paclitaxel and carboplatin in the first-line metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. The participants has histologically or cytologically confirmed Non-Small Cell Lung Cancer (NSCLC)Stage IIIB with effusion. Mixed Non-Small Cell Lung Cancer (NSCLC) tumors will be categorized by the predominant cell type. Primary or metastatic site may be used for histology
2. For squamous cell histology or for centrally located mediastinal masses (< 3 cm from the carina) identified by computed tomography scan (CT) or chest x-ray, the participant must undergo a magnetic resonance imaging (MRI) of the chest or I.V. contrast CT scan within 3 weeks of randomization, to exclude major airway or blood vessel invasion (in the investigator's opinion) by cancer
3. The participant has measurable disease (Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
4. The participant's Eastern Cooperative Oncology Group (ECOG) performance status is 0-1
5. The participant's age at the time of study entry is ≥ 18 years
6. The participant has adequate hematologic function as defined by an absolute neutrophil count (ANC) ≥ 1500/μL, hemoglobin ≥ 9.5 g/dL, and a platelet count ≥ 100,000/μL obtained within 2 weeks prior to randomization
7. The participant has adequate hepatic function as defined by a total bilirubin ≤ 1.5 mg/dL, and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 × the upper limit of normal (ULN), or ≤ 5 × the ULN in the presence of known liver metastases)
8. The participant has adequate renal function as defined by serum creatinine ≤ 1.5 × the institutional ULN. If creatinine is above the ULN, the patient's creatinine clearance (CrCl) is ≥ 60 mL/min
9. The participant has urinary protein ≤ 1+ on dipstick or routine urinalysis; if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine for protein must demonstrate < 1 g of protein in 24 hours to allow participation
10. The participant has adequate coagulation function, as defined by international normalized ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 5 seconds above ULN if not receiving anticoagulation therapy. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin, have therapeutic INR, no active bleeding (defined as within 14 days randomization) and no pathological condition that carries a high risk of bleeding (eg, tumor involving major vessels or known varices)
11. Because the teratogenicity of Olaratumab is not known, women of childbearing potential (WOCBP) and sexually active males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to randomization and for the duration of study participation
12. The participant has resolution to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4 (NCI-CTCAE v 4.02) of all clinically significant toxic effects of prior locoregional therapy, surgery, chemoembolization, or other anticancer therapy. The exceptions for such effects are events that pertain to the lab values found elsewhere in these inclusion criteria. (For example, criterion # 6 states that a patient with hemoglobin ≥ 9.5 g/dL is considered eligible, even though NCI-CTCAE v 4.02 defines this value as Grade 2 anemia.)
13. The participant has a life expectancy of ≥ 3 months
14. The participant has provided signed informed consent

Exclusion Criteria:

1. The participant has untreated central nervous system (CNS) metastases. Participants are eligible if they are clinically stable, off all steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, stereotactic radiosurgery)ending at least 2 weeks prior to randomization, or after surgical resection performed at least 4 weeks prior to randomization
2. The participant has radiologically documented evidence of major blood vessel invasion or encasement by cancer, or of intratumor cavitation
3. The participant received prior systemic chemotherapy or biologic therapy (eg erlotinib) for Stage IIIB/IV NSCLC outside of the adjuvant setting. Participants who received prior cytotoxic chemotherapy or biologic therapy in the adjuvant setting will not be excluded based on such therapy
4. The participant has a history of another primary cancer, with the exception of a) curatively resected nonmelanomatous skin cancer b) curatively treated cervical carcinoma in situ c)other primary solid tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years prior to randomization
5. The participant is receiving concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemo-embolization, targeted therapy, or an investigational agent
6. The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
7. The participant has an uncontrolled thrombotic or hemorrhagic disorder
8. The participant has a history of gross hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon) within 2 months of randomization
9. The participant has a serious non-healing wound, ulcer, or bone fracture within 28 days prior to randomization
10. The participant has undergone major surgery within 28 days prior to randomization
11. The participant has received adjuvant chemotherapy 21 days prior to randomization or has participated in clinical trials of experimental agents within 28 days prior to randomization
12. The participant has an elective or a planned major surgery to be performed during the course of the trial
13. The participant has peripheral neuropathy ≥ Grade 2 NCI-CTCAE v 4.02
14. The participant has known human immunodeficiency virus (HIV) positivity
15. The participant, if female, is pregnant or lactating
16. The participant has received previous therapy with any agent that targets platelet derived growth factor (PDGF) or platelet derived growth factor receptor (PDGFR)
17. The participant has a known allergy to any of the treatment components
18. The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to that of Olaratumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (20):
  - ImClone Investigational Site, Birmingham, Alabama
  - ImClone Investigational Site, Bakersfield, California
  - ImClone Investigational Site, Highland, California
  - ImClone Investigational Site, Stamford, Connecticut
  - ImClone Investigational Site, Port Saint Lucie, Florida
  - ImClone Investigational Site, Joliet, Illinois
  - ImClone Investigational Site, Baton Rouge, Louisiana
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Charlotte, North Carolina
  - ImClone Investigational Site, Gastonia, North Carolina
  - ImClone Investigational Site, Huntersville, North Carolina
  - ImClone Investigational Site, Canton, Ohio
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Massillon, Ohio
  - ImClone Investigational Site, Portland, Oregon
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Round Rock, Texas
  - ImClone Investigational Site, Temple, Texas
  - ImClone Investigational Site, Madison, Wisconsin
- Canada (2):
  - ImClone Investigational Site, Calgary, Alberta
  - ImClone Investigational Site, Edmonton, Alberta

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had evidence of progressive disease (PD), died or crossover to Olaratumab were considered to have completed the study.
Groups:
- Olaratumab + Paclitaxel + Carboplatin: Olaratumab: 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, administered IV at 25mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel 200 milligram/square meter (mg/m2) over 3 hrs (Day 1) Carboplatin Area Under Concentration (AUC)=6 (Day 1) of each 21-day cycle
  Paclitaxel 200 mg/m2 over 3 hrs (Day 1) Carboplatin AUC=6 (Day 1) of each 21-day cycle
  Participants who experience progressive disease may cross over to olaratumab monotherapy.
  Paclitaxel: 200 mg/m2 is then administered intravenously (IV) over 3 hours
  carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
- Crossover to Olaratumab Monotherapy: Olaratumab was administered IV at 15 mg/kg on Day 1 and Day 8 every 3 weeks.
Period: Treatment With or Without Olaratumab
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab Monotherapy
Started | 70 | 67 | 0
Received at Least 1 Dose of Study Drug | 67 | 64 | 0
Death Due to Any Cause | 53 | 47 | 0
Alive/On Study at End/Off Treatment | 11 | 10 | 0
Completed | 64 | 57 | 0
Not Completed | 6 | 10 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0
Not completed — Other Therapy Started | 2 | 1 | 0
Not completed — Never Treated/Death | 1 | 0 | 0
Period: Crossover to Olaratumab Monotherapy
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab Monotherapy
Started | 0 | 0 | 18 (18 participants who had progressive disease crossed over to monotherapy.)
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All phase 2 participants who were randomized and received any dose of study drug.
Groups:
- Olaratumab + Paclitaxel + Carboplatin: Olaratumab 15 mg/kg over 30 mins (Days 1 and 8) plus Paclitaxel 200 mg/m2 over 3 hrs (Day 1) Carboplatin AUC=6 (Day 1) of each 21-day cycle
  Participants can remain on study after completing chemotherapy and receive olaratumab monotherapy on Days 1 and 8, provided there is ongoing evidence of clinical benefit.
  Olaratumab: 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, administered IV at 25mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel: 200 mg/m2 is then administered IV over 3 hours
  Carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
- Total: Total of all reporting groups
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.77) | 63.8 (9.67) | 63.7 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 40 | 34 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 64 | 62 | 126
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 6 | 16
  White | 54 | 56 | 110
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participants] — ECOG performance status classified participants according to their functional impairment. Scores ranged from 0 (fully active) to 5 (death).
  participants
    ECOG PS 0 | 25 | 16 | 41
    ECOG PS 1 | 42 | 48 | 90
Stratification Factor Case Report Form (CRF) [Number; unit: participants]
  Non-Squamous Cell Carcinoma | 48 | 48 | 96
  Squamous Cell Carcinoma | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the day of randomization to the first evidence of progression by RECIST version 1.1, or death from any cause. Participants who died without a reported prior progression were considered to have progressed on the day of their death. Participants who did not progress and were subsequently lost to follow-up had their data censored at the day of their last tumor assessment. If there was no radiologic assessment at baseline or post baseline, participants were censored at the date of randomization. If death or progressive disease (PD) occurred after 2 or more consecutive missing radiographic visits, censoring occurred at the date of the last radiographic visit prior to the missed visits.
Time Frame: Baseline to Measured PD or Death From Any Cause (Up to 31 Months)
Population: All randomized participants who received any dose of study drug. Participants censored: paclitaxel + carboplatin = 13, olaratumab + paclitaxel + carboplatin = 20, and crossover to olaratumab = 4. 1 participant did not cross over to Olaratumab until after efficacy data completion, no efficacy data collected on this participant.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Olaratumab + Paclitaxel + Carboplatin: Olaratumab: 15 mg/kg of Olaratumab on Days 1 and 8 of each 21-day cycle, administered IV at 25mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel: 200 mg/m2 is then administered IV over 3 hours
  Carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
- Crossover to Olaratumab: Olaratumab monotherapy administered on Days 1 and 8 of each 21-day cycle.
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab
Number analyzed (Participants) | 67 | 64 | 17
weeks | 19.1 [16.4 to 23.6] | 19.0 [15.3 to 25] | 8.3 [5.0 to 13.4]
Statistical Analysis 1: Comparison: Olaratumab + Paclitaxel + Carboplatin vs Crossover to Olaratumab; Test type: Superiority or Other; p = 0.2133, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.86 to 1.93]

2. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to Study Completion (Up to 43 Months)
Population: All randomized participants who received any dose of study drug. 1 participant did not cross over to Olaratumab until after efficacy data completion, no efficacy data collected on this participant.
Measure: Number; unit: participants
Groups:
- Olaratumab + Pacilitaxel + Carboplatin: Olaratumab: 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, administered IV at 25mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel: 200 mg/m2 is then administered IV over 3 hours
  Carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
Arm/Group | Olaratumab + Pacilitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab
Number analyzed (Participants) | 67 | 64 | 17
participants
  AE | 66 | 63 | 10
  SAE's | 30 | 21 | 2

3. Secondary Outcome: Safety and Tolerability of Olaratumab Administered at a More Rapid Rate (25mg/Min With Minimum Infusion Time of 30 Minutes), Determined by Number of Participants With Treatment Related Adverse Events
Time Frame: Up to 43 Months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab
Number analyzed (Participants) | 67 | 64 | 17
participants
  AE | 66 | 63 | 10
  SAE's | 30 | 21 | 2

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from date of randomization to the date of death from any cause. If the participant is alive at the end of the follow-up period or is lost to follow-up, OS was censored on the last date the participants is known to be alive.
Time Frame: Baseline to Death From Any Cause (Up to 31 Months)
Population: All randomized participants who received any dose of study drug. OS data was not analyzed in the crossover olaratumab arm. Participants censored: olaratumab + paclitaxel + carboplatin = 19 and paclitaxel + carboplatin = 20.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 67 | 64
weeks | 51.3 [39.7 to 68.7] | 50.1 [41.4 to 75.9]
Statistical Analysis 1: Comparison: Olaratumab + Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.8731, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.68 to 1.57]

5. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) Objective Tumor Response Rate (ORR)
Description: The ORR is equal to the percentage of participants achieving a best overall response of partial response or complete response (PR + CR), according to RECIST version 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions; PD was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir; Stable Disease (SD) was defined as small changes that did not meet above criteria. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR/total number of participants)*100.
Time Frame: Baseline to Measured PD or Study Discontinuation (Up to 31 Months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab
Number analyzed (Participants) | 67 | 64 | 17
percentage of participants | 41.8 [29.8 to 54.5] | 34.4 [22.9 to 47.3] | 0 [0.0 to 19.5]
Statistical Analysis 1: Comparison: Olaratumab + Paclitaxel + Carboplatin; Test type: Superiority or Other; p = 0.4721, Fisher Exact

6. Secondary Outcome: Median Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are first met for Complete Response (CR)/Partial Response (PR) (whichever is first recorded) until the first date that the criteria for PD are met (taking as a reference for PD the smallest measurement recorded since the treatment started), initiation of other/additional antitumor therapy is first reported, or death, is objectively documented.
Time Frame: First Criteria Met for CR or PR to Measured PD Start of Other Antitumor Therapy or Death From Any Cause (Up to 31 Months)
Population: All randomized participants who received any dose of study drug and had achieved tumor response of CR or PR. Median Duration of Response data was not analyzed in the crossover olaratumab arm.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin
Number analyzed (Participants) | 28 | 22
weeks | 14.4 [12.7 to 18.1] | 12.9 [11.4 to 35.0]

7. Secondary Outcome: Pharmacodynamics of Olaratumab
Description: Pharmacodynamics of Olaratumab was determined by analysis of pharmacodynamic markers vascular endothelial growth factor (VEGF) and platelet derived growth factor (PDGF).
Time Frame: Cycle 1: Days 1, 8, and 15 pre- and post-infusion of Olaratumab; Cycles 2-6: day 1 only, pre- and post-infusion of Olaratumab
Population: No data was available due to the collection of plasma samples was not fit for the assessment of PDGFs, as the collection procedure did not prevent platelet activation resulting in elevated levels of PDGFs in the circulation. Pharmacodynamics data was not analyzed in the paclitaxel + carboplatin arm or the crossover to olaratumab arm.
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Participants With Anti-Olaratumab Antibodies
Description: Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Baseline to Study Completion (Up to 8 Months)
Population: All randomized participants who had baseline and post baseline Anti-Olaratumab antibodies. Those participants who did not meet eligibility criteria were not included in this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Crossover to Olaratumab
Number analyzed (Participants) | 45 | 4
percentage of participants | 4.4 | 0.0

9. Secondary Outcome: Pharmacokinetics (PK) - Area Under the Curve (AUC) 0-168 of Olaratumab
Description: AUC(0-168) = area under the concentration versus time curve from time zero to 168 hours post dose.
Time Frame: Cycle 3, Day 1: Predose, 30 minutes (min), 1.5 hours (hrs), 24,48,96,168 Hrs Post Dose
Population: All randomized participants who received any dose of study drug and had evaluable PK data in Cycle 3. PK data was not analyzed in the paclitaxel + carboplatin arm or the crossover to olaratumab arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (ug*hr/mL)
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6
microgram*hour/milliliter (ug*hr/mL) | 47600 (29.2)

10. Secondary Outcome: PK - Maximum Concentration (Cmax) of Olaratumab
Time Frame: Cycle 3, Day 1: Predose, 30 min, 1.5 hrs, 24,48,96,168 Hrs Post Dose
Population: All randomized participants who received any dose of study drug and had evaluable PK data in Cycle 3 first dose. PK data was not analyzed in the paclitaxel + carboplatin arm or the crossover to olaratumab arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (ug/mL)
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6
micrograms/milliliter (ug/mL) | 489 (13)

11. Secondary Outcome: PK - Half-Life (t1/2) of Olaratumab
Time Frame: Cycle 3, Day 1: Predose, 30 min, 1.5 hrs, 24,48,96,168 Hrs Post Dose
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: days
Groups:
- Olaratumab + Paclitaxel + Carboplatin: Olaratumab: 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, administered IV at 25 mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel: 200 mg/m2 is then administered IV over 3 hours
  Carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6
days | 5.79 [4.29 to 8.78]

12. Secondary Outcome: PK - Clearance (Cl) of Olaratumab
Time Frame: Cycle 3, Day 1: Predose, 30 min, 1.5 hr, 24,48,96,168 Hrs Post Dose
Population: All randomized participants who received any dose of study drug and had evaluable PK data in Cycle 3 first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6
Liter/hour (L/h) | 0.0218 (24.8)

13. Secondary Outcome: PK - Steady State Volume of Distribution (Vss) of Olaratumab
Time Frame: Cycle 3, Day 1: Predose, 30 min, 1.5 hrs, 24,48,96,168 Hrs Post Dose
Population: All randomized participants who received any dose of study drug and had evaluable PK data in Cycle 3 first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Olaratumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6
Liter (L) | 4.22 (9.51)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Olaratumab + Paclitaxel + Carboplatin: Olaratumab 15 mg/kg over 30 mins (Days 1 and 8) plus Paclitaxel 200 mg/m2 over 3 hrs (Day 1) Carboplatin AUC=6 (Day 1) of each 21-day cycle
  Participants can remain on study after completing chemotherapy and receive olaratumab monotherapy on Days 1 and 8, provided there is ongoing evidence of clinical benefit.
  Olaratumab: 15 mg/kg of IMC-3G3 on Days 1 and 8 of each 21-day cycle, administered IV at 25mg/min, with a minimum infusion time of 30 minutes.
  Paclitaxel: 200 mg/m2 is then administered IV over 3 hours
  Carboplatin: AUC=6 administered IV over 30 minutes on Day 1 of each 3-week cycle for a maximum of six cycles. Once the maximum of 6 cycles of carboplatin are reached the participant may continue on olaratumab maintenance for up to 12 months.
Arm/Group | Olaratumab + Paclitaxel + Carboplatin | Paclitaxel + Carboplatin | Crossover to Olaratumab
Serious Adverse Events (participants affected / at risk) | 30/67 | 21/64 | 3/18
Other Adverse Events (participants affected / at risk) | 67/67 | 64/64 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Paclitaxel + Carboplatin (N=67) | Paclitaxel + Carboplatin (N=64) | Crossover to Olaratumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incorrect drug administration duration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olaratumab + Paclitaxel + Carboplatin (N=67) | Paclitaxel + Carboplatin (N=64) | Crossover to Olaratumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 23 (45) | 26 (41) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 15 (32) | 6 (19) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 8 (19) | 4 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 29 (67) | 18 (39) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (64) | 15 (32) | 0 (0)
Vision blurred (Eye disorders) | 5 (6) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (8) | 4 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 24 (29) | 27 (29) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 29 (47) | 19 (26) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 11 (14) | 7 (9) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 34 (57) | 35 (47) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 16 (16) | 8 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 28 (36) | 22 (30) | 1 (1)
Asthenia (General disorders) | 4 (5) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 4 (4) | 2 (2) | 0 (0)
Chills (General disorders) | 8 (8) | 6 (6) | 1 (1)
Fatigue (General disorders) | 43 (75) | 33 (49) | 3 (4)
Infusion related reaction (General disorders) | 6 (7) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 12 (15) | 5 (5) | 0 (0)
Pain (General disorders) | 4 (4) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 6 (8) | 5 (8) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (8) | 5 (5) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 4 (4) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 4 (4) | 5 (8) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 12 (17) | 1 (2)
White blood cell count decreased (Investigations) | 4 (4) | 2 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 28 (35) | 12 (16) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 10 (11) | 11 (15) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (10) | 5 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 9 (14) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (17) | 11 (13) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (43) | 14 (24) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 12 (15) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (7) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (11) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (18) | 15 (21) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 16 (20) | 3 (3)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 10 (17) | 13 (15) | 3 (3)
Dysgeusia (Nervous system disorders) | 13 (13) | 9 (10) | 1 (1)
Headache (Nervous system disorders) | 13 (14) | 10 (14) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 23 (33) | 17 (29) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (5) | 4 (5) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (39) | 22 (38) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (6) | 6 (6) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (19) | 12 (12) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2/27 (2) | 0/30 (0) | 0/8 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (9) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 13 (16) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 6 (9) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 37 (45) | 38 (40) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 6 (9) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 6 (7) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (5) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days